CLINICAL TRIAL: NCT06601686
Title: Neuromodulation-assisted Ego-disengagement: The NEURO-EGO Study
Brief Title: Neuromodulation-assisted Ego-disengagement: The NEURO-EGO Study Stage 1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Tiny Blue Dot Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2023-0613; A535100 (Other: UW Madison); Protocol Version 10/9/25 (Other: UW Madison)
Record Dates: First submitted 2024-09-10; First posted 2024-09-19 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Healthy
Keywords: meditation; brain stimulation
MeSH Terms: interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Masking Description: Participants will not know whether they receive sham or real stimulation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Stimulation (Experimental): Participants will undergo sham, TES or TES-TI stimulation while completing cognitive assessments.
  Interventions: Device: Transcranial electrical stimulation (TES); Device: Transcranial electrical stimulation with temporal interference (TES-TI); Device: Sham stimulation

INTERVENTIONS:
Device: Transcranial electrical stimulation (TES) — TES uses specific electrode arrangement patterns to selectively stimulate the brain. Participants will wear an hdEEG (high density electroencephalography) cap which will allow intermittent periods of stimulation from TES.
Device: Transcranial electrical stimulation with temporal interference (TES-TI) — TES-TI uses specific electrode arrangement patterns to selectively stimulate the brain. Participants will wear an hdEEG (high density electroencephalography) cap which will allow intermittent periods of stimulation from TES-TI.
Device: Sham stimulation — TES-TI sham includes receiving stimulation from all electrodes at the same frequency. Sham TES will include administration of transcranial random noise stimulation (tRNS), random oscillating current. It will also include periods with no stimulation and a ramping up period followed by no stimulation.

SUMMARY:
The goal of this clinical trial is to learn whether brain stimulation technology can help people reach a meditative state quickly and easily without years of meditation training. The researchers want to see if this will help people distance themselves from their thoughts and feeling, and if this will lead to improvements in openness and wellbeing the same way meditation can.

Participants will:

* Complete questionnaires
* Perform a guided meditation task (The Bell Task)
* Wear a high density electrocochleography (hdEEG) cap
* Undergo brain stimulation
* Perform cognitive tasks

DETAILED DESCRIPTION:
This study is being done to evaluate the relative effectiveness of distinct types of non-invasive brain stimulation - NIBS (TES-TI and TES) on subjective ego disengagement and cortical activity in experienced meditators.

Phase 1 (registered to this record) involves administering 2 distinct types of deep brain stimulation techniques to a small sample (N=12) of experienced meditators to determine which type of neuromodulation, when focused on disruption of posteromedial cortex (PMC) activity, most robustly facilitates positive ego-disengagement compared to sham; and to discern the region of the PMC where disruption is most effective in achieving ego disengagement.

Phase 2 (registered to a separate record, NCT06601699) will use the most effective stimulation and PMC parameters to meditation naïve healthy adults.

ELIGIBILITY:
Inclusion Criteria:

* Adults, ages 18 to 80 of any identified gender
* Medically healthy
* English-speaking (able to provide consent and complete questionnaires)
* Healthy adults with a consistent meditation practice
* Citizen or legal resident

Exclusion Criteria:

* Any current or past history of neurological disorders or acquired neurological disease (e.g. stroke, traumatic brain injury), including intracranial lesions
* Any current or past history of bipolar disorder and/or hypomania
* Any current or past history of psychosis
* History of head trauma resulting in prolonged loss of consciousness; or a history of greater than 3 grade I concussions
* Current history of poorly controlled headaches including intractable or poorly controlled migraines
* Any systemic illness or unstable medical condition that may cause a medical emergency in case of a provoked seizure (cardiac malformation, cardiac dysrhythmia, asthma, etc.)
* History of fainting spells of unknown or undetermined etiology that might constitute seizures
* History of seizures, diagnosis of epilepsy, history of abnormal (epileptiform) EEG, or family history of treatment resistant epilepsy with the exception of a single seizure of benign etiology (e.g. febrile seizures) in the judgment of a board-certified neurologist
* Possible pregnancy. All female participants of child-bearing age are required to have a pregnancy test
* Any metal in the brain, skull or head
* Any contraindications to MRI
* Any medical devices or implants (i.e. cardiac pacemaker, medication infusion pump, cochlear implant, vagal nerve stimulator, dental implants (this includes a permanent retainer)) unless otherwise approved by the responsible MD
* Substance abuse or dependence within the past six months
* Any medication that may alter seizure threshold i.e., ADHD stimulants (Adderall, amphetamine); Tricyclic/atypical antidepressants (Amitriptyline, Dioxepine, Imipramine Maprotiline, Nortriptyline, Bupropion); Antipsychotics (Chlorpromazine, Clozapine), Bronchodilators (theophylline, aminophylline); Antibiotics (fluoroquinolones, imipenem, penicillin, cephalosporins, metronidazole, isoniazid); Antiviral (Valacyclovir, Ritonavir); OTC (Diphenhydramine)
* Claustrophobia (a fear of small or closed places)
* Back problems that would prevent lying flat for up to two hours
* Motion sickness
* Any hair braid, dreadlocks, hair pieces, or extensions which cannot be taken out or adjusted to permit comfortable and comprehensive participation before the MRI scans and/or stimulation sessions
* Any head coverings or headdress that participant feels uncomfortable removing for the purposes of the MRI scans and/or stimulation session

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2026-10 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
Ego-Disengagement scale | Data collected at one study visit (anytime up to 2 weeks on study)
  Ego-disengagement will be measured using the bell task. This meditation task consists of five "bell trials." During each trial, subjects will be asked to focus on the sound of a bell until it fades, then on the space left empty by the faded sound, resting free from thoughts as long as possible (meditation condition). Afterward, subjects will respond to a few questions designed to assess their level of ego-disengagement during the trials. This is a five-question form that asks subjects to rate, on a scale from 0-4, the degree to which they were perceiving something, imagining something, thinking about themselves, or thinking about something during the previous bell trial and then to rate the valence of their emotional state during the trial from 1 (highly negative) to 6 (highly positive).
Cortical activity - change in gamma band power | Data collected at one study visit (anytime up to 2 weeks on study)
  Gamma band power will be measured with hdEEG during stimulation. A decrease indicates greater level of ego disengagement.
Cortical activity - change in alpha band power | Data collected at one study visit (anytime up to 2 weeks on study)
  Alpha band power will be measured with hdEEG during stimulation. An increase indicates greater level of ego disengagement.

SECONDARY OUTCOMES:
Change in Big Five Aspects Scale (BFAS) | baseline to follow up (up to 6 weeks)
  This is a 44-item inventory that measures five different personality traits by asking subjects to respond to various items (e.g., I see myself as someone who is talkative) on a scale from 1 (disagree strongly) to 5 (agree strongly).
Change in Fulfilled Life Scale (FLS) | baseline to follow up (up to 6 weeks)
  This is a 32-item inventory that asks subjects to respond to various items (e.g., When I look back on my life, I feel deep inner contentment) on a scale from 1 (does not apply at all) to 6 (applies completely) and is designed to assess subjects' feelings of having lived a full life.
Change in PROMIS Anxiety | baseline to follow up (up to 6 weeks)
  This is an 8-item inventory asking subjects to rate from 1-5 the frequency with which they have experienced components of anxiety in the last seven days. Higher scores reflect greater anxiety.
Change in PROMIS Depression | baseline to follow up (up to 6 weeks)
  This is an 8-item inventory asking subjects to rate from 1-5 the frequency with which they have experienced components of depression in the last seven days. Higher scores reflect greater depression.
Change in Perceived Stress Scale (PSS) | baseline to follow up (up to 6 weeks)
  This is a 10-item inventory asking subjects to rate from 0-4 the frequency with which they have felt various kinds of stress in the last month. Participants rate each item on a scale ranging from "Never (0)" to "Very often (4)". Seven of the items with positive statements are scored in reverse. As the scores obtained from the scale increase, the perceived stress level of the person increases. Scores range from 0-40.
Change in Questionnaire for Eudaimonic Well-Being (QEWB) | baseline to follow up (up to 6 weeks)
  This is a 21-item inventory asking subjects to rate from 0-4 the extent to which they agree with various statements designed to assess their overall well-being. Scores range from 0-84 with higher scores indicating higher levels of well-being.
Change in Psychological Wellbeing Scale (PWB) | baseline to follow up (up to 6 weeks)
  The PWB Scale is a tool designed to measure various aspects of an individual's psychological well-being. The scale consists of 18 items and assesses six key dimensions of well-being: Autonomy - The ability to make independent decisions and resist social pressures; Environmental Mastery -The capacity to manage one's life and surrounding environment effectively; Personal Growth - A sense of continued development and realization of one's potential; Positive Relations with Others -The presence of meaningful, trusting relationships; Purpose in Life - Having goals and a sense of direction in life; Self-Acceptance - A positive attitude towards oneself and one's past life. There are three items per each dimension. Each item is rated on a scale from 1 (strongly disagree) to 7 (strongly agree), higher scores indicate higher wellbeing.
Change in IQSS Flourishing Measure | baseline to follow up (up to 6 weeks)
  The Human Flourishing Measures is designed to assess various domains of human well-being and flourishing. Developed by the Human Flourishing Program at Harvard University, this measure aims to provide a comprehensive understanding of an individual's overall well-being, across different domains such as, health, life satisfaction, purpose, close relationships. The questionnaire consists of 12 items, rated from 0 (Strongly disagree) to 10 (Strongly agree). High scores imply that people perceive themselves very positively in terms of human flourishing.
Change in Metacognitive Processes of Decentering Scale (MPoD) | baseline to follow up (up to 6 weeks)
  The MPoD is designed to measure the ability to decenter from internal experiences. Decentering involves viewing thoughts and feelings as temporary and objective events in the mind, rather than as reflections of the self. Items are scored from 1 (never or very rarely) to 5 (very often or always) for a total range of scores from 15-75 where higher scores indicate higher levels of engagement with trait-like metacognitive processes of decentering.
Change in Experiences Questionnaire (EQ) | baseline to follow up (up to 6 weeks)
  This 20-item self-report measure assesses trait levels of decentering and rumination. Decentering refers to the ability to view one's thoughts and feelings as temporary, objective events rather than reflections of the self. It is a key component of mindfulness and is often developed through meditation practices. The component Rumination includes items that measure the tendency to dwell on negative thoughts and feelings. For example, items might ask about the frequency of repetitive, negative thinking. Items are scored from 1 (never) to 5 (all the time) where higher scores indicate indicate higher decentering and rumination.
Change in Self-Reflection Insight Scale (SRIS) | baseline to follow up (up to 6 weeks)
  The SRIS is a psychometric tool designed to measure two critical components of self-awareness: self-reflection and insight. It provides a reliable means of assessing individuals' tendencies to engage in introspection and their ability to gain clear understanding from such introspection. Participants respond to each item using a Likert scale ranging from 1 (strongly disagree) to 6 (strongly agree). Higher scores indicate self-awareness.
Change in Non-Attachment Scale (NAS) | baseline to follow up (up to 6 weeks)
  NAS is designed to assess the extent to which individuals experience nonattachment in their daily lives. The NAS consists of 30 items that participants rate based on their agreement from 1 (strongly disagree) to 6 (strongly agree). The items are designed to capture various aspects of nonattachment, such as the ability to let go of thoughts and emotions, and the tendency to experience life without excessive clinging or aversion. Higher scores indicate more non-attachment.
Change in Non-Attachment to Self Scale (NTS) | baseline to follow up (up to 6 weeks)
  NTS is a psychological measure designed to assess the degree to which individuals are not fixated on self-related concepts, thoughts, and feelings. It captures the ability to interact with these self-related elements flexibly and without trying to control them. It is a single factor, 7-item scale, where each item is scored from 1 (Strongly Disagree) to 7 (Strongly Agree). Higher scores indicate more non-attachment to self.
Change in Five Facet Mindfulness Questionnaire (FFMQ) | baseline to follow up (up to 6 weeks)
  FFMQ is a comprehensive self-report instrument designed to assess mindfulness across five distinct dimensions. The FFMQ consists of 39 items, divided into five subscales, each representing a different facet of mindfulness: observing, describing, acting with awareness, nonjudging of inner experience, nonreactivity to inner experience. Participants respond to each item using a Likert scale ranging from 1 (never or very rarely true) to 5 (very often or always true). Higher scores on the FFMQ reflects a higher level of mindfulness (a better outcome).
Change in Drexel Defusion Scale (DDS) | baseline to follow up (up to 6 weeks)
  DDS is a psychometric instrument developed to measure the construct of defusion, which refers to the ability to achieve psychological distance from internal experiences such as thoughts and feelings. Participants respond to each item using a six-point Likert scale ranging from 0 (not at all) to 5 (very much), for a total possible range of scores from 0-50, higher scores indicate increased ability to defuse.
Change in Relationship Questionnaire (RQ) | baseline to follow up (up to 6 weeks)
  RQ is a self-report instrument designed to assess various dimensions of interpersonal relationship styles. The RQ consists of 4 items, each describing a specific relationship style. Participants rate each item on a 7-point Likert scale, ranging from "1 = Strongly Disagree" to "7 = Strongly Agree."
Change in UCLA Loneliness Scale (ULS) | baseline to follow up (up to 6 weeks)
  ULS is a widely used tool designed to measure an individual's subjective feelings of loneliness and social isolation. The scale consists of 20 items. Each item is rated on a 4-point Likert scale ranging from 1 (Never) to 4 (Often). Some items are reverse-scored to control for response bias. The total score ranges from 20 to 80, with higher scores indicating greater levels of loneliness.
Change in Social Connectedness Scale (SCS) | baseline to follow up (up to 6 weeks)
  SCS, developed by Richard M. Lee and Steven B. Robbins in 1995, is a self-report questionnaire designed to measure the extent to which individuals feel connected to others in their social environment. The scale assesses feelings of closeness and belongingness, which are crucial for psychological well-being. The scale consists of 20 items. Each item is rated on a Likert scale ranging from 1 (strongly disagree) to 6 (strongly agree). Higher scores indicate a greater sense of social connectedness, while lower scores suggest feelings of social isolation or disconnection.
Change in Attachment Style Questionnaire (ASQ) | baseline to follow up (up to 6 weeks)
  ASQ is a self-report measure designed to assess adult attachment styles. This questionnaire helps identify how individuals typically think, feel, and behave in close relationships. The ASQ consists of 40 items rated on 6-point Likert Scale (1 Totally disagree - 6 Totally Agree). It measures five dimensions of attachment, that is, confidence, discomfort with closeness, need for approval, preoccupation with relationship, relationship as secondary.
Change in Emotional Intelligence Scale (EIS) | baseline to follow up (up to 6 weeks)
  EIS is designed to measure the ability to identify, assess, and manage the emotions of oneself, others, and groups. The EIS consists of 33 items. Participants rate each item on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Higher scores indicate higher emotional intelligence.
Change in Barratt Impulsiveness Scale (BIS-11) | baseline to follow up (up to 6 weeks)
  BIS-11 is a widely used self-report measure designed to assess the personality/behavioral construct of impulsiveness. The BIS-11 consists of 30 items, each rated on a 4-point Likert scale ranging from 1 (rarely/never) to 4 (almost always/always).
  The BIS-11 measures three primary dimensions of impulsiveness:
  1. Attentional Impulsiveness: Difficulty focusing attention and a tendency to make quick decisions.
  2. Motor Impulsiveness: Acting on the spur of the moment and a lack of perseverance.
  3. Non-Planning Impulsiveness: A lack of forethought or consideration of future consequences.
  Each of these dimensions is further broken down into subscales, providing a detailed profile of an individual's impulsivity traits. The total score ranges from 30 to 120, with higher scores indicating higher levels of impulsiveness.
Change in Dickman Impulsivity Inventory (DII) | baseline to follow up (up to 6 weeks)
  DII is a self-report measure designed to assess two distinct types of impulsivity: functional impulsivity and dysfunctional impulsivity. Functional Impulsivity is characterized by the tendency to act quickly and effectively in situations where such behavior is beneficial.
  Dysfunctional Impulsivity involves acting with less forethought than most people, leading to negative outcomes. The DII consists of 23 items that are true or false statements. Each true statement is scored as 1. The scores for each subscale (functional impulsivity and dysfunctional impulsivity) are summed, with higher scores indicating higher levels of functional or dysfunctional impulsivity.
Change in Vividness of Visual Imagery Questionnaire (VVIQ) | baseline to follow up (up to 6 weeks)
  VVIQ is a tool developed to assess the vividness of an individual's visual imagination. Items are scored on a 5-point Likert Scale from 1 (no image at all) to 5 (Perfectly clear and as vivid as normal vision). The questionnaire includes scenarios such as visualizing a friend's face, a rising sun, and other common scenes to gauge the vividness of the mental images. Higher scores indicate more vivid visual imagery.
Implicit Association Task: Response Time | Data collected at one study visit (anytime up to 2 weeks on study)
  IAT is a psychological tool designed to measure the strength of automatic associations between mental representations of objects or concepts. The IAT typically involves categorizing words or images that appear on a computer screen into different groups as quickly as possible. For example, participants might be asked to categorize words as either "pleasant" or "unpleasant" and images as either "young" or "old." The speed at which participants categorize the items is crucial. Faster response times indicate stronger implicit associations between the categories being tested.
Implicit Association Task: Accuracy Reported as the Number of Misclassifications | Data collected at one study visit (anytime up to 2 weeks on study)
  IAT is a psychological tool designed to measure the strength of automatic associations between mental representations of objects or concepts. The IAT typically involves categorizing words or images that appear on a computer screen into different groups as quickly as possible. For example, participants might be asked to categorize words as either "pleasant" or "unpleasant" and images as either "young" or "old." Participants complete 8 blocks of 24 trials each, consisting of two groups of 4 incongruent and 4 congruent blocks. Within each group of blocks, the first trial serves as a practice trial.
Implicit Association Task: D-Score | Data collected at one study visit (anytime up to 2 weeks on study)
  IAT is a psychological tool designed to measure the strength of automatic associations between mental representations of objects or concepts. The IAT typically involves categorizing words or images that appear on a computer screen into different groups as quickly as possible. For example, participants might be asked to categorize words as either "pleasant" or "unpleasant" and images as either "young" or "old."
  Reported here is the the D-score that measures the standardized difference between the average response times for congruent and incongruent pairings, adjusted for the number of errors. It typically ranges from -2 to 2. A score near zero indicates selfless processing of fear. Positive scores are expected to represent identification with fear. Conversely, negative scores are expected to represent negative self-referential evaluation of fear.
Rapid Discrimination Task: Speed | Data collected at one study visit (anytime up to 2 weeks on study)
  The Rapid Discrimination Task is a cognitive task used to assess an individual's ability to quickly and accurately distinguish between different stimuli. Participants are presented with a series of stimuli, which can vary in attributes such as shape, color, size, or emotional expression. The task requires participants to make quick decisions about the stimuli, often under time constraints.
  Both the speed and accuracy of responses are measured to assess perceptual and cognitive abilities. For the Rapid Discrimination Task, two black and white geometric shapes one next to the other are presented using Eprime. In some slides, the two shapes will be identical and in others they will differ by one line or outside edge of the shape being slightly different than the other. The participant is instructed to press the 'S' button on the keyboard if they are the same or the 'L' button if they are different. This will repeat for up to 25 minutes until the task ends.
Rapid Discrimination Task: Accuracy | Data collected at one study visit (anytime up to 2 weeks on study)
  The Rapid Discrimination Task is a cognitive task used to assess an individual's ability to quickly and accurately distinguish between different stimuli. Participants are presented with a series of stimuli, which can vary in attributes such as shape, color, size, or emotional expression. The task requires participants to make quick decisions about the stimuli, often under time constraints.
  Both the speed and accuracy of responses are measured to assess perceptual and cognitive abilities. For the Rapid Discrimination Task, two black and white geometric shapes one next to the other are presented using Eprime. In some slides, the two shapes will be identical and in others they will differ by one line or outside edge of the shape being slightly different than the other. The participant is instructed to press the 'S' button on the keyboard if they are the same or the 'L' button if they are different. This will repeat for up to 25 minutes until the task ends.
Spontaneous Mentation Task | Data collected at one study visit (anytime up to 2 weeks on study)
  Participants with eyes open or closed will be prompted by a beep to report the last thing that was going through their mind (image, thought, feeling, emotion …) just before the sound. After this open-ended report, participants will also be asked to rate on a VAS scale (e.g., from 0 to 5) their awareness, some quality aspects of their mentation content (e.g, how thought-like or image-like it was; or the degree of cognitive effort).
  [will the VAS score be reported?]
Automatic Emotion Regulation Task | Data collected at one hour MRI visit (scheduled within 2 weeks on study)
  The automatic emotion regulation (AER) task is designed to investigate how individuals modulate their emotional responses without conscious effort. In this task, participants are exposed to various emotional stimuli, in this experiment image, which are typically categorized as positive (e.g., a puppy or a sunset), negative (e.g., the image of a natural disaster or of a person in distress), or neutral (e.g., the photo of a chair or of a building). These stimuli are presented rapidly to minimize conscious regulation efforts.
  During the task, functional MRI data will be recorded. The goal is to measure how effectively participants can automatically regulate their emotional reactions. Data analysis focuses on comparing responses across different emotional conditions to infer the efficiency of automatic emotion regulation.
  Participants will rate on a VAS scale (from 1 to 10) the intensity of the emotional content evoked by each picture, higher numbers are more intense.
Resting State Task | Data collected at one hour MRI visit (scheduled within 2 weeks on study)
  Participants are simply asked to rest quietly, awake but relaxed, to record brain activity without any external stimuli influencing it.
  The signal measured within each voxel is based on the blood-oxygen-level-dependent (BOLD) contrast, which reflects changes in blood flow and oxygenation associated with neural activity.
  While resting state activity can help the interpretation of different task states, it will be mainly evaluated as a measure in itself to assess baseline brain functional organization of the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Melanie Boly, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Neuromodulation-assisted Ego-disengagement: the NEURO-EGO Study Stage 2 — https://clinicaltrials.gov/study/NCT06601699